CLINICAL TRIAL: NCT00567567
Title: Phase III Randomized Trial of Single vs. Tandem Myeloablative Consolidation Therapy for High-Risk Neuroblastoma
Brief Title: Comparing Two Different Myeloablation Therapies in Treating Young Patients Who Are Undergoing a Stem Cell Transplant for High-Risk Neuroblastoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ANBL0532; NCI-2009-01065 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000576571; 08-524; COG-ANBL0532; ANBL0532 (Other: Childrens Oncology Group); ANBL0532 (Other: CTEP); U10CA180886 (NIH); U10CA098543 (NIH)
Record Dates: First submitted 2007-12-04; First posted 2007-12-05 (Estimated); Results first posted 2017-06-27 (Actual); Last update posted 2022-04-28 (Actual); Status verified 2021-12

CONDITIONS: Localized Resectable Neuroblastoma; Localized Unresectable Neuroblastoma; Recurrent Neuroblastoma; Regional Neuroblastoma; Stage 4 Neuroblastoma; Stage 4S Neuroblastoma
MeSH Terms: conditions — Neuroblastoma | interventions — Carboplatin; Cisplatin; 1,2-diaminocyclohexaneplatinum II citrate; Platinum; Cyclophosphamide; Doxorubicin; Etoposide; Filgrastim; Granulocyte Colony-Stimulating Factor; Isotretinoin; Melphalan; Peripheral Blood Stem Cell Transplantation; Thiotepa; Topotecan; Vincristine

ARMS (2):
- Consolidation Arm A: single myeloablative consolidation (Active Comparator): Patients receive melphalan IV over 15-30 minutes on days -7 to -5, etoposide IV over 24 hours and carboplatin IV over 24 hours on days -7 to -4, and G-CSF SC or IV beginning on day 0 and continuing until blood counts recover. Patients undergo autologous PBSCT on day 0.
  Interventions: Procedure: Autologous Hematopoietic Stem Cell Transplantation; Drug: Carboplatin; Drug: Cisplatin; Drug: Cyclophosphamide; Drug: Doxorubicin Hydrochloride; Drug: Etoposide; Radiation: External Beam Radiation Therapy; Biological: Filgrastim; Drug: Isotretinoin; Other: Laboratory Biomarker Analysis; Drug: Melphalan; Procedure: Peripheral Blood Stem Cell Transplantation; Other: Pharmacological Study; Drug: Topotecan Hydrochloride; Drug: Vincristine Sulfate Liposome
- Consolidation Arm B: tandem myeloablative consolidation (Experimental): Patients receive thiotepa IV over 2 hours on days -7 to -5, cyclophosphamide IV over 1 hour on days -5 to -2, and G-CSF SC or IV beginning on day 0 and continuing until blood counts recover. Following clinical recovery from initial myeloablative therapy, patients also receive melphalan, etoposide, and carboplatin as in Arm A. Patients undergo autologous PBSCT on day 0.
  Interventions: Procedure: Autologous Hematopoietic Stem Cell Transplantation; Drug: Carboplatin; Drug: Cisplatin; Drug: Cyclophosphamide; Drug: Doxorubicin Hydrochloride; Drug: Etoposide; Radiation: External Beam Radiation Therapy; Biological: Filgrastim; Drug: Isotretinoin; Other: Laboratory Biomarker Analysis; Drug: Melphalan; Procedure: Peripheral Blood Stem Cell Transplantation; Other: Pharmacological Study; Drug: Thiotepa; Drug: Topotecan Hydrochloride; Drug: Vincristine Sulfate Liposome

INTERVENTIONS:
Procedure: Autologous Hematopoietic Stem Cell Transplantation — Undergo autologous peripheral blood stem cell transplant
  Other Names: Autologous Hematopoietic Cell Transplantation; autologous stem cell transplantation
Drug: Carboplatin — Given IV
  Other Names: Blastocarb; Carboplat; Carboplatin Hexal; Carboplatino; Carbosin; Carbosol; Carbotec; CBDCA; Displata; Ercar; JM-8; Nealorin; Novoplatinum; Paraplatin; Paraplatin AQ; Paraplatine; Platinwas; Ribocarbo
Drug: Cisplatin — Given IV
  Other Names: Abiplatin; Blastolem; Briplatin; CDDP; Cis-diammine-dichloroplatinum; Cis-diamminedichloridoplatinum; Cis-diamminedichloro Platinum (II); Cis-diamminedichloroplatinum; Cis-dichloroammine Platinum (II); Cis-platinous Diamine Dichloride; Cis-platinum; Cis-platinum II; Cis-platinum II Diamine Dichloride; Cismaplat; Cisplatina; Cisplatinum; Cisplatyl; Citoplatino; Citosin; Cysplatyna; DDP; Lederplatin; Metaplatin; Neoplatin; Peyrone's Chloride; Peyrone's Salt; Placis; Plastistil; Platamine; Platiblastin; Platiblastin-S; Platinex; Platinol; Platinol- AQ; Platinol-AQ; Platinol-AQ VHA Plus; Platinoxan; Platinum; Platinum Diamminodichloride; Platiran; Platistin; Platosin
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR- 138719
Drug: Doxorubicin Hydrochloride — Given IV
  Other Names: 5,12-Naphthacenedione, 10-[(3-amino-2,3,6-trideoxy-alpha-L-lyxo-hexopyranosyl)oxy]-7,8, 9,10-tetrahydro-6,8,11-trihydroxy-8-(hydroxyacetyl)-1-methoxy-, hydrochloride, (8S-cis)- (9CI); ADM; Adriacin; Adriamycin; Adriamycin Hydrochloride; Adriamycin PFS; Adriamycin RDF; ADRIAMYCIN, HYDROCHLORIDE; Adriamycine; Adriblastina; Adriblastine; Adrimedac; Chloridrato de Doxorrubicina; DOX; DOXO-CELL; Doxolem; Doxorubicin.HCl; Doxorubin; Farmiblastina; FI 106; FI-106; hydroxydaunorubicin; Rubex
Drug: Etoposide — Given IV
  Other Names: Demethyl Epipodophyllotoxin Ethylidine Glucoside; EPEG; Lastet; Toposar; Vepesid; VP 16-213; VP-16; VP-16-213
Radiation: External Beam Radiation Therapy — Undergo EBRT
  Other Names: Definitive Radiation Therapy; EBRT; External Beam Radiotherapy; External Beam RT; external radiation; External Radiation Therapy; external-beam radiation
Biological: Filgrastim — Given IV or SC
  Other Names: FILGRASTIM, LICENSE HOLDER UNSPECIFIED; G-CSF; Neupogen; r-metHuG-CSF; Recombinant Methionyl Human Granulocyte Colony Stimulating Factor; rG-CSF; Tevagrastim
Drug: Isotretinoin — Given orally
  Other Names: 13-cis retinoic acid; 13-cis-Retinoate; 13-cis-Retinoic Acid; 13-cis-Vitamin A Acid; 13-cRA; Accure; Accutane; Amnesteem; cis-Retinoic Acid; Cistane; Claravis; Isotretinoinum; Isotrex; Isotrexin; Neovitamin A; Neovitamin A Acid; Oratane; Retinoicacid-13-cis; Ro 4-3780; Ro-4-3780; Roaccutan; Roaccutane; Roacutan; Sotret
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Melphalan — Given IV
  Other Names: Alanine Nitrogen Mustard; CB-3025; L-PAM; L-Phenylalanine Mustard; L-sarcolysin; L-Sarcolysin Phenylalanine mustard; L-Sarcolysine; Melphalanum; Phenylalanine Mustard; Phenylalanine nitrogen mustard; Sarcoclorin; Sarkolysin; WR-19813
Procedure: Peripheral Blood Stem Cell Transplantation — Undergo autologous peripheral blood stem cell transplant
  Other Names: PBPC transplantation; PBSCT; Peripheral Blood Progenitor Cell Transplantation; Peripheral Stem Cell Support; Peripheral Stem Cell Transplant; Peripheral Stem Cell Transplantation
Other: Pharmacological Study — Correlative studies
Drug: Thiotepa — Given IV
  Other Names: 1,1',1''-Phosphinothioylidynetrisaziridine; Girostan; N,N', N''-Triethylenethiophosphoramide; Oncotiotepa; STEPA; Tepadina; TESPA; Tespamin; Tespamine; Thio-Tepa; Thiofosfamide; Thiofozil; Thiophosphamide; Thiophosphoramide; Thiotef; Tifosyl; TIO TEF; Tio-tef; Triethylene thiophosphoramide; Triethylenethiophosphoramide; Tris(1-aziridinyl)phosphine sulfide; TSPA; WR 45312
  Arms: Consolidation Arm B: tandem myeloablative consolidation
Drug: Topotecan Hydrochloride — Given IV
  Other Names: Hycamptamine; Hycamtin; SKF S-104864-A; Topotecan HCl; topotecan hydrochloride (oral)
Drug: Vincristine Sulfate Liposome — Given IV
  Other Names: Marqibo

SUMMARY:
This randomized phase III trial compares two different high-dose chemotherapy regimens followed by a stem cell transplant in treating younger patients with high-risk neuroblastoma. Drugs used in chemotherapy work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving combination chemotherapy before surgery may make the tumor smaller and reduce the amount of normal tissue that needs to be removed. Giving these treatments before a peripheral blood stem cell transplant helps kill any tumor cells that are in the body and helps make room in the patient?s bone marrow for new blood-forming cells (stem cells) to grow. After treatment, stem cells are collected from the patient's blood and stored. High-dose chemotherapy and radiation therapy is then given to prepare the bone marrow for the stem cell transplant. The stem cells are then returned to the patient to replace the blood-forming cells that were destroyed by the high- chemotherapy. It is not yet known which regimen of high-dose chemotherapy is more effective for patients with high-risk neuroblastoma undergoing a peripheral blood stem cell transplant.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To improve the 3-year event-free survival (EFS) rate of high-risk neuroblastoma patients through treatment with a tandem consolidation of thiotepa/cyclophosphamide followed by carboplatin/etoposide/melphalan (CEM) as compared to single CEM consolidation.

II. To improve the rate of end-induction complete response and very good partial response, compared to historical controls, by use of a topotecan-containing induction regimen.

III. To improve the 3-year local control rate, compared to historical controls, by increasing the local dose of radiation to the residual primary tumor for patients with less than a gross total resection.

SECONDARY OBJECTIVES:

I. To evaluate the pharmacogenetic relationship of cyclophosphamide metabolizing enzymes (CYP2B6, CYP2C9, and GSTA1 genotypes) with toxicity and response following dose-intensive cyclophosphamide and topotecan induction chemotherapy.

II. To determine if resection completeness is predictive of a) local control rate; or b) EFS rate in patients with high-risk neuroblastoma.

III. To prospectively describe the complications related to efforts at local control (surgery and radiation therapy) in patients with high-risk neuroblastoma.

IV. To describe the neurologic outcome of patients with paraspinal primary neuroblastoma tumors.

V. To determine the variability of 13-cis-retinoic-acid pharmacokinetics and relationship to pharmacogenomic parameters and determine if pharmacokinetics and/or genetic variations correlate with EFS or systemic toxicity as follows: a) To determine the variability of 13-cis-retinoic-acid pharmacokinetics and relationship to pharmacogenomic parameters. b) To determine if 13-cis-retinoic-acid pharmacokinetic levels are predictive of the EFS rate or associated with systemic toxicity following 13-cis-retinoic acid. c) To determine if pharmacogenomic variations are predictive of the EFS rate or associated with systemic toxicity following 13-cis-retinoic acid.

VI. To evaluate total topotecan pharmacokinetics and correlate with patient specific data for use in an ongoing topotecan population pharmacokinetic analysis.

VII. To evaluate the presence and function of T cells capable of recognizing neuroblastoma by assessing: a) if T cells recognizing the neuroblastoma antigen, survivin, circulate at diagnosis; b) if these T cells can be expanded using autologous antigen presenting cells (APCs); c) if these T cells will kill neuroblastoma cells as detected in functional assays; and d) if the presence and activity of anti-neuroblastoma immunity is decreased by stem cell transplantation.

VIII. To characterize the recovery of T- cell numbers after myeloablative consolidation and hematopoietic stem cell transplant (HSCT) and assess the impact of tandem myeloablative consolidation on T- cell recovery.

IX. To characterize minimal residual disease burden using reverse transcriptase-polymerase chain reaction (RT-PCR) evaluation of a panel of neuroblastoma specific transcripts in patient bone marrow and peripheral blood following induction chemotherapy and after single versus tandem myeloablative chemotherapy and to evaluate impact on EFS.

X. To evaluate the EFS and overall survival (OS) rate for patients 12-18 months with Stage 4, MYCN nonamplified tumor with unfavorable histopathology or diploid DNA content or with indeterminant histology or ploidy and patients who are greater than 547 days of age with Stage 3, MYCN nonamplified tumor AND unfavorable histopathology or indeterminant histology following treatment with single myeloablative transplant.

OUTLINE:

INDUCTION CHEMOTHERAPY:

COURSES 1 AND 2: Patients receive cyclophosphamide IV over 30 minutes and topotecan hydrochloride IV over 30 minutes on days 1-5 and filgrastim (G-CSF) subcutaneously (SC) or IV beginning on day 6 and continuing until blood counts recover. Treatment repeats every 21 days for 2 courses. Patients undergo peripheral blood stem cell (PBSC) mobilization and harvest after course 2.

COURSES 3 AND 5: Patients receive cisplatin IV over 1 hour on days 1-4, etoposide IV over 1 hour on days 1-3, and G-CSF SC or IV beginning on day 5 and continuing until blood counts recover. Treatment repeats every 21 days for 2 courses. Patients undergo surgical resection of soft tissue disease after course 5 (or after course 6 if medically necessary).

COURSES 4 AND 6: Patients receive cyclophosphamide IV over 6 hours on days 1-2, doxorubicin hydrochloride IV over 24 hours on days 1-3, vincristine IV on days 1-3, and G-CSF SC or IV beginning on day 5 and continuing until blood counts recover. Treatment repeats every 21 days for 2 courses.

Patients are then stratified by initial stage of disease and MYCN status, biologic characteristics, and response to induction chemotherapy (complete response/very good partial response vs partial response vs mixed response/no response). Patients are randomized to 1 of 2 arms. Patients 12?18 months old (i.e., 365-547 days) with stage IV, MYCN nonamplified tumor with unfavorable histopathology or diploid DNA content or with indeterminant histology or ploidy AND patients who are 547 days of age with stage III, MYCN nonamplified tumor AND unfavorable histopathology or indeterminant histology will be nonrandomly assigned to Arm A. Patients begin consolidation chemotherapy no later than 8 weeks after the start of induction course 6.

CONSOLIDATION THERAPY:

ARM A (single myeloablative consolidation): Patients receive melphalan IV over 15-30 minutes on days -7 to -5, etoposide IV over 24 hours and carboplatin IV over 24 hours on days -7 to -4, and G-CSF SC or IV beginning on day 0 and continuing until blood counts recover. Patients undergo autologous peripheral blood stem cell transplant (PBSCT) on day 0.

ARM B (tandem myeloablative consolidation): Patients receive thiotepa IV over 2 hours on days -7 to -5, cyclophosphamide IV over 1 hour on days -5 to -2, and G-CSF SC or IV beginning on day 0 and continuing until blood counts recover. Following clinical recovery from initial myeloablative therapy, patients also receive melphalan, etoposide, and carboplatin as in Arm A. Patients undergo autologous PBSCT on day 0.

RADIOTHERAPY: Patients undergo external beam radiation therapy (EBRT) to primary site of disease as well as to MIBG-avid sites seen at pre-transplantation (i.e., end-induction) evaluation between 28-42 days post-transplant. Additional radiotherapy is administered to residual tumor at primary site.

MAINTENANCE THERAPY: Patients are encouraged to enroll onto Children?s Oncology Group (COG)-ANBL0032 following assessment of tumor response after completion of the consolidation phase and radiotherapy. Beginning on day 60 post-transplantation patients receive oral isotretinoin twice daily on days 1-14. Treatment repeats every 28 days for up to 6 months in the absence of disease progression or unacceptable toxicity. Patients undergo blood and tissue sample collection periodically for the following analyses; correlation between peak serum concentration level and the existence of polymorphisms, event-free survival, and toxicity rates; pharmacogenomics for uridine diphosphate (UDP) glucuronosyltransferase 1 family, polypeptide A1 (UGT1A1), UGT2B7, CYP2C8 and CYP3A7 alleles; topotecan systemic clearance; survivin-specific cytotoxic T-lymphocytes (CTLs) detected using peptide/major histocompatibility complex (MHC) tetramers in human leukocyte antigen (HLA)-A2+ patients; interferon (IFN)-gamma production in enzyme-linked immunospot (ELISPOT) assays to APCs loaded with tumor ribonucleic acid (RNA), survivin RNA, or control RNA; response of APC-stimulated CTL response to neuroblastoma cells; rate of T cell recovery; and proportion of patients with neuroblastoma detected in bone marrow and peripheral blood using RT-PCR and immunohistochemistry (IHC).

After completion of study treatment, patients are followed up periodically for 5 years and then annually for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of neuroblastoma or ganglioneuroblastoma by histology or as evidenced by the presence of clumps of tumor cells in bone marrow and elevated catecholamine metabolites in urine meeting any of the following criteria:

  * Patients with newly diagnosed neuroblastoma with International Neuroblastoma Staging System (INSS) stage 4 disease are eligible with the following:

    * MYCN amplification (i.e., greater than four-fold increase in MYCN signals as compared to reference signals), regardless of age or additional biologic features
    * Age > 18 months (i.e., > 547 days) regardless of biologic features
    * Age 12-18 months (i.e., 365-547 days) with none of the following three favorable biologic features (i.e., non-amplified MYCN, favorable pathology, and deoxyribonucleic acid [DNA] index > 1)
  * Patients with newly diagnosed neuroblastoma with INSS stage 3 are eligible with the following:

    * MYCN amplification (i.e., greater than four-fold increase in MYCN signals as compared to reference signals), regardless of age or additional biologic features
    * Age > 18 months (i.e., > 547 days) with unfavorable pathology, regardless of MYCN status
  * Patients with newly diagnosed INSS stage 2a or 2b with MYCN amplification (i.e., greater than four-fold increase in MYCN signals as compared to reference signals), regardless of age or additional biologic features
  * Patients with newly diagnosed INSS stage 4s with MYCN amplification (i.e., greater than four-fold increase in MYCN signals as compared to reference signals), regardless of additional biologic features
  * Patients >= 365 days initially diagnosed with INSS stage 1, 2, or 4S and who progressed to a stage 4 without interval chemotherapy

    * Must have been enrolled on COG-ANBL00B1
* Creatinine clearance or radioisotope glomerular filtration rate ? 70mL/min OR serum creatinine based on age/gender as follows:

  * 1 month to < 6 months: 0.4 mg/dL
  * 6 months to < 1 year: 0.5 mg/dL
  * 1 to < 2 years: 0.6 mg/dL
  * 2 to < 6 years: 0.8 mg/dL
  * 6 to < 10 years: 1 mg/dL
  * 10 to < 13 years: 1.2 mg/dL
  * 10 to < 16 years: 1.5 mg/dL (male), 1.4 mg/dL (female)
  * >= 16 years: 1.7 mg/dL (male), 1.4 mg/dL (female)
* Total bilirubin ? 1.5 times upper limit of normal (ULN) for age
* Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) < 10 times ULN for age
* Not pregnant or nursing
* Negative pregnancy test
* Shortening fraction >= 27% by echocardiogram (ECHO) OR left ventricular ejection fraction (LVEF) >= 50% by radionuclide angiogram
* No known contraindication (e.g., size, weight or physical condition) to peripheral blood stem cell collection
* No prior systemic therapy except for localized emergency radiation to sites of life-threatening or function-threatening disease
* No more than one course of chemotherapy per low- or intermediate-risk neuroblastoma therapy prior to determination of MYCN amplification and histology

Max Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 665 (Actual)
Dates: Start 2007-11-05 (Actual); Primary Completion 2015-02-27 (Actual); Study Completion 2022-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julie R Park, Principal Investigator — Children's Oncology Group
Locations (190):
- United States (169):
  - Children's Hospital of Alabama, Birmingham, Alabama
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - USA Health Strada Patient Care Center, Mobile, Alabama
  - Phoenix Childrens Hospital, Phoenix, Arizona
  - The University of Arizona Medical Center-University Campus, Tucson, Arizona
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Kaiser Permanente Downey Medical Center, Downey, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Loma Linda University Medical Center, Loma Linda, California
  - Miller Children's and Women's Hospital Long Beach, Long Beach, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - Valley Children's Hospital, Madera, California
  - Children's Hospital and Research Center at Oakland, Oakland, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Children's Hospital of Orange County, Orange, California
  - Lucile Packard Children's Hospital Stanford University, Palo Alto, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Rady Children's Hospital - San Diego, San Diego, California
  - UCSF Medical Center-Mount Zion, San Francisco, California
  - UCSF Medical Center-Parnassus, San Francisco, California
  - Harbor-University of California at Los Angeles Medical Center, Torrance, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Rocky Mountain Hospital for Children-Presbyterian Saint Luke's Medical Center, Denver, Colorado
  - University of Connecticut, Farmington, Connecticut
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Alfred I duPont Hospital for Children, Wilmington, Delaware
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Broward Health Medical Center, Fort Lauderdale, Florida
  - Lee Memorial Health System, Fort Myers, Florida
  - Golisano Children's Hospital of Southwest Florida, Fort Myers, Florida
  - University of Florida Health Science Center - Gainesville, Gainesville, Florida
  - Memorial Regional Hospital/Joe DiMaggio Children's Hospital, Hollywood, Florida
  - Nemours Children's Clinic-Jacksonville, Jacksonville, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - Nicklaus Children's Hospital, Miami, Florida
  - Florida Hospital Orlando, Orlando, Florida
  - Nemours Children's Clinic - Orlando, Orlando, Florida
  - UF Cancer Center at Orlando Health, Orlando, Florida
  - Nemours Children's Clinic - Pensacola, Pensacola, Florida
  - Sacred Heart Hospital, Pensacola, Florida
  - Johns Hopkins All Children's Hospital, St. Petersburg, Florida
  - Saint Joseph's Hospital/Children's Hospital-Tampa, Tampa, Florida
  - Saint Mary's Hospital, West Palm Beach, Florida
  - Children's Healthcare of Atlanta - Egleston, Atlanta, Georgia
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Augusta University Medical Center, Augusta, Georgia
  - Memorial Health University Medical Center, Savannah, Georgia
  - Lurie Children's Hospital-Chicago, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Saint Jude Midwest Affiliate, Peoria, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Riley Hospital for Children, Indianapolis, Indiana
  - Saint Vincent Hospital and Health Care Center, Indianapolis, Indiana
  - Blank Children's Hospital, Des Moines, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - University of Kansas Cancer Center, Kansas City, Kansas
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Norton Children's Hospital, Louisville, Kentucky
  - Tulane University Health Sciences Center, New Orleans, Louisiana
  - Children's Hospital New Orleans, New Orleans, Louisiana
  - Eastern Maine Medical Center, Bangor, Maine
  - Maine Children's Cancer Program, Scarborough, Maine
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Floating Hospital for Children at Tufts Medical Center, Boston, Massachusetts
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Massachusetts Medical School, Worcester, Massachusetts
  - C S Mott Children's Hospital, Ann Arbor, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Ascension Saint John Hospital, Detroit, Michigan
  - Michigan State University Clinical Center, East Lansing, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Helen DeVos Children's Hospital at Spectrum Health, Grand Rapids, Michigan
  - Spectrum Health at Butterworth Campus, Grand Rapids, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - Kalamazoo Center for Medical Studies, Kalamazoo, Michigan
  - Children's Hospitals and Clinics of Minnesota - Minneapolis, Minneapolis, Minnesota
  - University of Minnesota/Masonic Cancer Center, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - University of Missouri - Ellis Fischel, Columbia, Missouri
  - Children's Mercy Hospitals and Clinics, Kansas City, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Children's Hospital and Medical Center of Omaha, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Nevada Cancer Research Foundation CCOP, Las Vegas, Nevada
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Morristown Medical Center, Morristown, New Jersey
  - Saint Peter's University Hospital, New Brunswick, New Jersey
  - Rutgers Cancer Institute of New Jersey-Robert Wood Johnson University Hospital, New Brunswick, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - Saint Joseph's Regional Medical Center, Paterson, New Jersey
  - Overlook Hospital, Summit, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Albany Medical Center, Albany, New York
  - Brooklyn Hospital Center, Brooklyn, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - The Steven and Alexandra Cohen Children's Medical Center of New York, New Hyde Park, New York
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - Mount Sinai Hospital, New York, New York
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - University of Rochester, Rochester, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - New York Medical College, Valhalla, New York
  - Mission Hospital Inc-Memorial Campus, Asheville, North Carolina
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Novant Health Presbyterian Medical Center, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Rainbow Babies and Childrens Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Dayton Children's Hospital, Dayton, Ohio
  - The Toledo Hospital/Toledo Children's Hospital, Toledo, Ohio
  - Mercy Children's Hospital, Toledo, Ohio
  - University of Toledo, Toledo, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Legacy Emanuel Children's Hospital, Portland, Oregon
  - Legacy Emanuel Hospital and Health Center, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Lehigh Valley Hospital - Muhlenberg, Bethlehem, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Penn State Children's Hospital, Hershey, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Saint Christopher's Hospital for Children, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Prisma Health Richland Hospital, Columbia, South Carolina
  - BI-LO Charities Children's Cancer Center, Greenville, South Carolina
  - Greenville Cancer Treatment Center, Greenville, South Carolina
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - T C Thompson Children's Hospital, Chattanooga, Tennessee
  - East Tennessee Childrens Hospital, Knoxville, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - Dell Children's Medical Center of Central Texas, Austin, Texas
  - Driscoll Children's Hospital, Corpus Christi, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - Cook Children's Medical Center, Fort Worth, Texas
  - Covenant Children's Hospital, Lubbock, Texas
  - Methodist Children's Hospital of South Texas, San Antonio, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Primary Children's Hospital, Salt Lake City, Utah
  - University of Vermont and State Agricultural College, Burlington, Vermont
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Naval Medical Center - Portsmouth, Portsmouth, Virginia
  - Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia
  - Carilion Clinic Children's Hospital, Roanoke, Virginia
  - Seattle Children's Hospital, Seattle, Washington
  - Providence Sacred Heart Medical Center and Children's Hospital, Spokane, Washington
  - Madigan Army Medical Center, Tacoma, Washington
  - West Virginia University Charleston Division, Charleston, West Virginia
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin
- Australia (5):
  - The Children's Hospital at Westmead, Westmead, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Royal Brisbane and Women's Hospital, Herston, Queensland
  - Royal Children's Hospital-Brisbane, Herston, Queensland
  - Princess Margaret Hospital for Children, Perth, Western Australia
- Canada (13):
  - Alberta Children's Hospital, Calgary, Alberta
  - University of Alberta Hospital, Edmonton, Alberta
  - British Columbia Children's Hospital, Vancouver, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - IWK Health Centre, Halifax, Nova Scotia
  - McMaster Children's Hospital at Hamilton Health Sciences, Hamilton, Ontario
  - Kingston Health Sciences Centre, Kingston, Ontario
  - Children's Hospital, London, Ontario
  - Victoria Hospital, London, Ontario
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - Hospital for Sick Children, Toronto, Ontario
  - Centre Hospitalier Universitaire Sainte-Justine, Montreal, Quebec
  - Centre Hospitalier Universitaire de Quebec, Québec
- Starship Children's Hospital, Grafton, Auckland, New Zealand
- San Jorge Children's Hospital, San Juan, Puerto Rico
- Swiss Pediatric Oncology Group - Bern, Bern, Switzerland

REFERENCES:
- [Derived] Berko ER, Naranjo A, Daniels AA, McNulty SN, Krytska K, Druley T, Zelley K, Koneru B, Chen L, Polkosnik G, Irwin MS, Bagatell R, Maris JM, Reynolds CP, DuBois SG, Park JR, Mosse YP. Frequency and Clinical Significance of Clonal and Subclonal Driver Mutations in High-Risk Neuroblastoma at Diagnosis: A Children's Oncology Group Study. J Clin Oncol. 2025 May 10;43(14):1673-1684. doi: 10.1200/JCO-24-02407. Epub 2025 Mar 4. PMID 40036726
- [Derived] Liu KX, Naranjo A, Zhang FF, DuBois SG, Braunstein SE, Voss SD, Khanna G, London WB, Doski JJ, Geiger JD, Kreissman SG, Grupp SA, Diller LR, Park JR, Haas-Kogan DA. Prospective Evaluation of Radiation Dose Escalation in Patients With High-Risk Neuroblastoma and Gross Residual Disease After Surgery: A Report From the Children's Oncology Group ANBL0532 Study. J Clin Oncol. 2020 Aug 20;38(24):2741-2752. doi: 10.1200/JCO.19.03316. Epub 2020 Jun 12. PMID 32530765
- [Derived] Park JR, Kreissman SG, London WB, Naranjo A, Cohn SL, Hogarty MD, Tenney SC, Haas-Kogan D, Shaw PJ, Kraveka JM, Roberts SS, Geiger JD, Doski JJ, Voss SD, Maris JM, Grupp SA, Diller L. Effect of Tandem Autologous Stem Cell Transplant vs Single Transplant on Event-Free Survival in Patients With High-Risk Neuroblastoma: A Randomized Clinical Trial. JAMA. 2019 Aug 27;322(8):746-755. doi: 10.1001/jama.2019.11642. PMID 31454045
- See also: Data Available: Select individual patient-level data from this trial can be requested from the NCTN/NCORP Data Archive — https://nctn-data-archive.nci.nih.gov/

RESULTS

PARTICIPANT FLOW:
Groups:
- Single HST (CEM): Induction therapy + single myeloablative consolidation
- Tandem HST (CEM), Randomly Assigned: Induction therapy + tandem myeloablative consolidation
- Not Assigned: Patients that either failed during Induction therapy or refused randomization
Period: Overall Study
Arm/Group | Single HST (CEM) | Tandem HST (CEM), Randomly Assigned | Not Assigned
Started | 210 | 176 | 279
Completed | 58 | 42 | 1
Not Completed | 152 | 134 | 278
Not completed — Adverse Event | 0 | 2 | 5
Not completed — Death | 8 | 1 | 5
Not completed — Lack of Efficacy | 16 | 17 | 48
Not completed — Lost to Follow-up | 0 | 0 | 1
Not completed — Physician Decision | 16 | 18 | 84
Not completed — Withdrawal by Subject | 0 | 0 | 2
Not completed — Ineligible | 4 | 0 | 9
Not completed — Refusal by patient/parent/guardian | 9 | 16 | 122
Not completed — Enrolled another COG therapeutic study | 99 | 80 | 0
Not completed — Unable adequate stem cell for transplant | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Single HST (CEM) | Tandem HST (CEM), Randomly Assigned | Not Assigned | Total
Number analyzed (Participants) | 210 | 176 | 279 | 665
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 208 | 176 | 277 | 661
  Between 18 and 65 years | 2 | 0 | 2 | 4
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 3.2 (2.9) | 2.9 (2.4) | 3.4 (2.8) | 3.2 (2.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 95 | 78 | 118 | 291
  Male | 115 | 98 | 161 | 374
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 22 | 26 | 30 | 78
  Not Hispanic or Latino | 181 | 145 | 233 | 559
  Unknown or Not Reported | 7 | 5 | 16 | 28
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 1
  Asian | 8 | 5 | 10 | 23
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 3 | 4
  Black or African American | 23 | 18 | 40 | 81
  White | 157 | 132 | 203 | 492
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 20 | 21 | 23 | 64
Region of Enrollment [Number; unit: participants]
  New Zealand | 3 | 1 | 3 | 7
  Canada | 19 | 21 | 23 | 63
  United States | 176 | 146 | 243 | 565
  Australia | 11 | 8 | 10 | 29
  Switzerland | 1 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Event-free Survival Rate
Description: Comparison of EFS curves, starting from the time of randomization, by treatment group (single CEM vs. tandem CEM)
Time Frame: Three years, from time of randomization
Population: All eligible, randomized patients.
Measure: Number (95% Confidence Interval); unit: percent probability
Arm/Group | Single HST (CEM) | Tandem HST (CEM), Randomly Assigned
Number analyzed (Participants) | 179 | 176
percent probability | 48.8 [41.1 to 56.5] | 61.8 [53.8 to 69.8]
Statistical Analysis 1: Comparison: Single HST (CEM) vs Tandem HST (CEM), Randomly Assigned; The event-free survival distributions of patients randomized to Regimen A - Single HST (CEM) and randomized to Regimen B - Tandem HST (CEM) were compared using the log-rank test; Test type: Superiority or Other; p = 0.0082, Log Rank; Log Rank Test Statistic = 6.9883

2. Primary Outcome: Response After Induction Therapy
Description: Per the International Response Criteria: measurable tumor defined as product of longest x widest perpendicular diameter. Elevated catecholamine levels, tumor cell invasion of bone marrow also considered measurable tumor. Complete Response (CR)-no evidence of primary tumor or metastases. Very Good Partial Response (VGPR)->90% reduction of primary tumor; no metastases; no new bone lesions, all pre-existing lesions improved. Partial Response (PR)-50-90% reduction of primary tumor; >50% reduction in measurable sites of metastases; 0-1 bone marrow samples with tumor; number of positive bone sites decreased by >50%. Mixed Response (MR)->50% reduction of any measurable lesion (primary or metastases) with <50% reduction in other sites; no new lesions; <25% increase in any existing lesion. No Response (NR)-no new lesions; <50% reduction but <25% increase in any existing legions. Progressive Disease (PD)-any new/increased measurable lesion by >25%; previous negative marrow positive.
Time Frame: Study enrollment to the end of induction therapy
Population: Eligible patients evaluated for response at the end of induction therapy.
Measure: Number (95% Confidence Interval); unit: Proportion participants that responded
Arm/Group | Single HST (CEM) | Tandem HST (CEM), Randomly Assigned | Not Assigned
Number analyzed (Participants) | 206 | 176 | 233
Proportion participants that responded | 0.54 [0.47 to 0.61] | 0.48 [0.41 to 0.56] | 0.35 [0.29 to 0.41]
Statistical Analysis 1: Comparison: Single HST (CEM) vs Tandem HST (CEM), Randomly Assigned vs Not Assigned; Chi-square test of proportions in all patients to compare the proportion of responders (complete response [CR]+ very good partial response [VGPR]) at the end of induction therapy in this study to an analogous cohort of responders in A3973; Test type: Superiority or Other; p = 0.0034, Chi-squared; Chi-squared test statistic = 8.5751

3. Primary Outcome: Incidence Rate of Local Recurrence
Description: Cumulative incidence rate of local recurrence comparison between ANBL0532 patients randomized or assigned to receive single CEM transplant and boost radiation versus the historical A3973 patients who were transplanted and received boost radiation.
Time Frame: Up to 3 years
Population: Eligible patients randomized or assigned to the single HST (CEM) treatment arm who also received boost radiation.
Measure: Number (95% Confidence Interval); unit: Percentage 3-year cumulative incidence
Arm/Group | Single HST (CEM)
Number analyzed (Participants) | 77
Percentage 3-year cumulative incidence | 15.7 [7.5 to 23.9]
Statistical Analysis 1: Comparison: Single HST (CEM); The cumulative incidence rates of local recurrence between patients from ANBL0532 randomized or assigned to receive single CEM transplant and boost radiation and A3973 patients who were transplanted and received boost radiation were compared using Gray's test; Test type: Superiority or Other; p = 0.5615, Gray's test for competing risks; Gray's test statistic = 0.33709

4. Secondary Outcome: Duration of Greater Than or Equal to Grade 3 Neutropenia
Description: A logistic regression model will be used to test the ability of the number of days of neutropenia to predict the presence of a polymorphism.
Time Frame: Through completion of a participant's first cycle during induction, including treatment delays, assessed up to 39 days
Population: Eligible patients with available polymorphism and neutropenia toxicity data.
Measure: Median (Full Range); unit: Days
Arm/Group | Single HST (CEM) | Tandem HST (CEM), Randomly Assigned | Not Assigned
Number analyzed (Participants) | 117 | 103 | 129
Days | 7 [0 to 20] | 7 [0 to 39] | 7 [0 to 35]
Statistical Analysis 1: Comparison: Single HST (CEM) vs Tandem HST (CEM), Randomly Assigned vs Not Assigned; Test type: Superiority or Other; p = 0.0939, Regression, Logistic; Slope = -0.0557

5. Secondary Outcome: Duration of Greater Than or Equal to Grade 3 Thrombocytopenia
Description: A logistic regression model will be used to test the ability of the number of days of thrombocytopenia to predict the presence of a polymorphism.
Time Frame: Through completion of a participant's first cycle during induction, including treatment delays, assessed up to 46 days
Population: Eligible patients with available polymorphism and thrombocytopenia toxicity data.
Measure: Median (Full Range); unit: Days
Arm/Group | Single HST (CEM) | Tandem HST (CEM), Randomly Assigned | Not Assigned
Number analyzed (Participants) | 117 | 103 | 129
Days | 4 [0 to 30] | 4 [0 to 46] | 4 [0 to 44]
Statistical Analysis 1: Comparison: Single HST (CEM) vs Tandem HST (CEM), Randomly Assigned vs Not Assigned; Test type: Superiority or Other; p = 0.3277, Regression, Logistic; Slope = 0.0543

6. Secondary Outcome: Proportion of Patients With a Polymorphism
Description: A chi-square test will be used to test whether the response rate after two cycles of induction therapy and the presence of a polymorphism are independent in the study population.
Time Frame: Through completion of a participant's first two cycles during induction, including treatment delays, assessed up to 69 days
Population: Eligible patients with available polymorphism data and response data after two cycles of induction therapy. Measure value is the proportion of patients with a polymorphism.
Measure: Number; unit: Proportion of patients
Arm/Group | Single HST (CEM) | Tandem HST (CEM), Randomly Assigned | Not Assigned
Number analyzed (Participants) | 101 | 92 | 109
Proportion of patients | 0.96 | 0.96 | 0.97
Statistical Analysis 1: Comparison: Single HST (CEM) vs Tandem HST (CEM), Randomly Assigned vs Not Assigned; Null Hypothesis: The response rate after two cycles of induction therapy and the presence of a polymorphism are independent in the study population; Test type: Superiority or Other; p = 0.7598, Fisher Exact; Fisher's exact test was used instead of chi-square test due to small expected cell counts; Odds Ratio (OR) = 1.4328, 95% CI 2-sided [0.4105 to 5.001]

7. Secondary Outcome: Surgical Response
Description: Percentage of patients who achieved a surgical complete resection
Time Frame: Up to 3 years
Population: All eligible patients enrolled on ANBL0532.
Measure: Number; unit: Percentage of patients
Arm/Group | Single HST (CEM) | Tandem HST (CEM), Randomly Assigned | Not Assigned
Number analyzed (Participants) | 206 | 176 | 270
Percentage of patients | 83.98 | 84.09 | 58.89

8. Secondary Outcome: Type of Surgical or Radiotherapy Complication
Description: The Percentage of patients who experienced surgical or radiotherapy complications will be calculated. The complications are: bowel obstruction, chylous leaf, renal injury/atrophy/loss and diarrhea.
Time Frame: Up to 3 years
Population: All eligible patients enrolled on ANBL0532.
Measure: Number; unit: Percentage of patients
Arm/Group | Single HST (CEM) | Tandem HST (CEM), Randomly Assigned | Not Assigned
Number analyzed (Participants) | 206 | 176 | 270
Percentage of patients | 13.11 | 12.50 | 11.85

9. Secondary Outcome: Intraspinal Extension
Description: Percentage of patients with primary tumors with intraspinal extension.
Time Frame: Up to 5 years
Population: All eligible patients enrolled on ANBL0532.
Measure: Number; unit: Percentage of patients
Arm/Group | Single HST (CEM) | Tandem HST (CEM), Randomly Assigned | Not Assigned
Number analyzed (Participants) | 206 | 176 | 270
Percentage of patients | 8.25 | 9.66 | 7.78

10. Secondary Outcome: Peak Serum Concentration of Isotretinoin in Patients Enrolled on Either A3973, ANBL0032, ANBL0931, ANBL0532 and Future High Risk Studies
Description: Median peak serum concentration level of isotretinoin for patients enrolled on ANBL0532
Time Frame: Day 1 of each course
Population: Eligible patients evaluated for peak serum concentration level of isotretinoin.
Measure: Median (Full Range); unit: Micromolar
Arm/Group | Single HST (CEM) | Tandem HST (CEM), Randomly Assigned | Not Assigned
Number analyzed (Participants) | 91 | 76 | 49
Micromolar | 1.00 [0 to 9.22] | 1.36 [0 to 12.93] | 1.26 [0 to 11.78]
Statistical Analysis 1: Comparison: Single HST (CEM) vs Tandem HST (CEM), Randomly Assigned vs Not Assigned; The relationship between the peak serum isotretinoin concentration level with event-free survival was explored with a Cox proportional hazards model. Eligible patients treated with isotretinoin on A3973, ANBL0032, ANBL0532, or ANBL0931 with peak serum concentration level data were included in the analysis; Test type: Superiority or Other; p = 0.6853, Regression, Cox; Hazard Ratio (HR) = 1.015

11. Secondary Outcome: Pharmacogenetic Variants in Patients Enrolled on Either A3973, ANBL0032, ANBL0931, ANBL0532 and Future High Risk Studies
Description: To determine if pharmacogenomic variations are predictive of EFS, a logrank test comparison of patients with vs without a given polymorphism will be made. A Fisher's exact test will test for association of the presence of a polymorphism with the occurrence of systemic toxicity (CTC grade 3 or 4 skin, hypercalcemia, or hepatic toxicity). These tests will be performed for UGT1A1, UGT2B7, CYP2C8 and CYP3A7 alleles.
Time Frame: At baseline
Population: Data were not collected to assess this study aim.
Groups:
- All Patients: All eligible and evaluable patients enrolled on ANBL0532
Arm/Group | All Patients
Number analyzed (Participants) | 0

12. Secondary Outcome: Topotecan Systemic Clearance
Description: Median topotecan systemic clearance for courses 1 and 2.
Time Frame: Day 1 of courses 1-2
Population: Eligible patients evaluated for topotecan systemic clearance.
Measure: Median (Full Range); unit: L/h/m2
Arm/Group | Single HST (CEM) | Tandem HST (CEM), Randomly Assigned | Not Assigned
Number analyzed (Participants) | 82 | 76 | 103
L/h/m2 | 28.1 [14.9 to 49.4] | 28.1 [11.6 to 42.7] | 28.5 [16.3 to 54.7]

13. Secondary Outcome: Presence and Function of T Cells Capable of Recognizing Neuroblastoma
Time Frame: Up to 6 months (end of therapy)
Population: Data were not collected to assess this study aim.
Arm/Group | Single HST (CEM) | Tandem HST (CEM), Randomly Assigned | Not Assigned
Number analyzed (Participants) | 0 | 0 | 0

14. Secondary Outcome: Enumeration of Peripheral Blood Cluster of Differentiation (CD)3, CD4, and CD8 Cells
Description: A descriptive comparison of the median number of T-cells (CD3, CD4, CD8) between treatment arms (single vs. tandem myeloablative regimens) will be performed.
Time Frame: Up to 6 months after completion of assigned myeloablation therapy
Population: All eligible patients that had CD3, CD4 and CD8T-cell count evaluated at the end of reporting period 3.
Measure: Median (Full Range); unit: cells/mm^3
Arm/Group | Single HST (CEM) | Tandem HST (CEM), Randomly Assigned
Number analyzed (Participants) | 43 | 43
cells/mm^3
  CD3: number analyzed (Participants) | 43 | 42
  CD3 | 200 [23 to 1549] | 255.5 [13 to 2987]
  CD4: number analyzed (Participants) | 42 | 43
  CD4 | 73 [8 to 626] | 81 [4 to 1186]
  CD8: number analyzed (Participants) | 41 | 43
  CD8 | 104 [8 to 1170] | 151 [4 to 2529]

15. Secondary Outcome: Proportion of Patients With Neuroblastoma Detected in Bone Marrow and Peripheral Blood Using RT-PCR Technique
Description: Will be calculated overall and by treatment arm.
Time Frame: Baseline
Population: Data were not collected to assess this study aim.
Groups:
- All Eligible Patients: All Eligible Patients
Arm/Group | Single HST (CEM) | Tandem HST (CEM), Randomly Assigned | All Eligible Patients
Number analyzed (Participants) | 0 | 0 | 0

16. Secondary Outcome: EFS Pts Non-randomly Assigned to Single CEM (12-18 Mths, Stg. 4, MYCN Nonamplified Tumor/Unfavorable or Indeterminant Histopathology/Diploid DNA Content & Pts>547 Days, Stg.3, MYCN Nonamplified Tumor AND Unfavorable or Indeterminant Histopathology).
Description: Kaplan-Meier curves of EFS will be plotted, and the proportion of responders to induction therapy will be tabulated.
Time Frame: Up to 3 years
Population: All eligible patients non-randomly assigned to single CEM
Measure: Number (95% Confidence Interval); unit: percent probability
Arm/Group | Single HST (CEM)
Number analyzed (Participants) | 27
percent probability | 73.1 [55.1 to 91.2]

17. Secondary Outcome: OS in Patients 12-18 Months, Stage 4, MYCN Nonamplified Tumor/Unfavorable Histopathology/Diploid DNA Content/Indeterminant Histology/Ploidy and Patients > 547 Days, Stage 3, MYCN Nonamplified Tumor AND Unfavorable Histopathology/Indeterminant Histology
Description: Kaplan-Meier curves of OS will be plotted, and the proportion of responders to induction therapy will be tabulated.
Time Frame: Up to 3 years
Measure: Number (95% Confidence Interval); unit: percent probability
Arm/Group | Single HST (CEM)
Number analyzed (Participants) | 27
percent probability | 81.0 [65.1 to 96.9]

ADVERSE EVENTS:
Description: We've excluded the ineligibles from this table.
Arm/Group | Single HST (CEM) | Tandem HST (CEM), Randomly Assigned | Not Assigned
Serious Adverse Events (participants affected / at risk) | 16/206 | 15/176 | 12/269
Other Adverse Events (participants affected / at risk) | 196/206 | 163/176 | 230/269
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single HST (CEM) (N=206) | Tandem HST (CEM), Randomly Assigned (N=176) | Not Assigned (N=269)
13200-Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 2 (2)
17200-Blood and lymphatic system disorders - Other specify (Blood and lymphatic system disorders) | 0 (0) | 3 (3) | 0 (0)
25800-Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 1 (1)
33300-Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0)
39600-Hemolysis (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
39700-Hemolytic uremic syndrome (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
20000-Cardiac arrest (Cardiac disorders) | 3 (3) | 0 (0) | 1 (1)
51700-Left ventricular systolic dysfunction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
63100-Pericardial effusion (Cardiac disorders) | 1 (1) | 2 (2) | 2 (2)
72700-Right ventricular dysfunction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
31900-Eye disorders - Other specify (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
14900-Ascites (Gastrointestinal disorders) | 2 (2) | 2 (2) | 0 (0)
35900-Gastric hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
36700-Gastrointestinal disorders - Other specify (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
36900-Gastrointestinal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
53000-Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
55600-Mucositis oral (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0)
70100-Rectal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
75700-Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
81900-Typhlitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
82200-Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
24600-Death NOS (General disorders) | 0 (0) | 0 (0) | 2 (2)
37200-General disorders and administration site conditions - Other specify (General disorders) | 0 (0) | 1 (1) | 0 (0)
55700-Multi-organ failure (General disorders) | 4 (4) | 0 (0) | 2 (2)
40000-Hepatic failure (Hepatobiliary disorders) | 1 (1) | 1 (1) | 0 (0)
40600-Hepatobiliary disorders - Other specify (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
66500-Portal hypertension (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
66600-Portal vein thrombosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
20500-Catheter related infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
44800-Infections and infestations - Other specify (Infections and infestations) | 4 (4) | 0 (0) | 2 (2)
73700-Sepsis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
13800-Aortic injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
45400-Injury to inferior vena cava (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
47700-Intraoperative renal injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
10900-Activated partial thromboplastin time prolonged (Investigations) | 0 (0) | 1 (1) | 1 (1)
11600-Alanine aminotransferase increased (Investigations) | 3 (3) | 1 (1) | 2 (2)
15000-Aspartate aminotransferase increased (Investigations) | 3 (3) | 1 (1) | 3 (3)
17400-Blood bilirubin increased (Investigations) | 4 (4) | 1 (1) | 2 (2)
24100-Creatinine increased (Investigations) | 3 (3) | 0 (0) | 2 (2)
37500-GGT increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
45800-INR increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
58300-Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
65800-Platelet count decreased (Investigations) | 1 (1) | 0 (0) | 1 (1)
88200-Weight gain (Investigations) | 0 (0) | 1 (1) | 0 (0)
88500-White blood cell decreased (Investigations) | 1 (1) | 0 (0) | 1 (1)
41300-Hypercalcemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
41800-Hypernatremia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0)
42600-Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
42700-Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
43100-Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2)
43300-Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
43500-Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
54900-Metabolism and nutrition disorders - Other specify (Metabolism and nutrition disorders) | 1 (1) | 1 (3) | 0 (0)
81700-Tumor lysis syndrome (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
58000-Neoplasms benign malignant and unspecified (incl cysts and polyps) - Other specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
81200-Treatment related secondary malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0)
25300-Depressed level of consciousness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
29000-Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
56600-Myelitis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
58100-Nervous system disorders - Other specify (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
11100-Acute kidney injury (Renal and urinary disorders) | 3 (3) | 0 (0) | 3 (3)
71000-Renal and urinary disorders - Other specify (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
19200-Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
27800-Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
29700-Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
43900-Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (4) | 2 (2)
65900-Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 2 (2)
66300-Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
69000-Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
71500-Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 2 (2)
71600-Respiratory thoracic and mediastinal disorders - Other specify (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 1 (1)
75300-Skin ulceration (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
79000-Surgical and medical procedures - Other specify (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
42100-Hypertension (Vascular disorders) | 1 (1) | 1 (1) | 0 (0)
43600-Hypotension (Vascular disorders) | 1 (1) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single HST (CEM) (N=206) | Tandem HST (CEM), Randomly Assigned (N=176) | Not Assigned (N=269)
13200-Anemia (Blood and lymphatic system disorders) | 23 (35) | 22 (37) | 33 (42)
17200-Blood and lymphatic system disorders - Other specify (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
25800-Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 1 (1)
33300-Febrile neutropenia (Blood and lymphatic system disorders) | 32 (46) | 32 (41) | 46 (53)
20000-Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
20100-Cardiac disorders - Other specify (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
39000-Heart failure (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
63100-Pericardial effusion (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
72700-Right ventricular dysfunction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
27900-Ear and labyrinth disorders - Other specify (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
38900-Hearing impaired (Ear and labyrinth disorders) | 6 (6) | 4 (4) | 3 (3)
11200-Adrenal insufficiency (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1)
31900-Eye disorders - Other specify (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
10100-Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
10300-Abdominal pain (Gastrointestinal disorders) | 5 (5) | 5 (8) | 6 (6)
14900-Ascites (Gastrointestinal disorders) | 2 (2) | 3 (3) | 0 (0)
22100-Colitis (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (1)
25700-Diarrhea (Gastrointestinal disorders) | 20 (21) | 7 (7) | 10 (10)
26600-Duodenal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
29400-Enterocolitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
31200-Esophagitis (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (2)
36400-Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
36700-Gastrointestinal disorders - Other specify (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
44200-Ileal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
44600-Ileus (Gastrointestinal disorders) | 2 (2) | 0 (0) | 8 (8)
46300-Intra-abdominal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
53000-Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
55600-Mucositis oral (Gastrointestinal disorders) | 20 (21) | 16 (16) | 6 (6)
57600-Nausea (Gastrointestinal disorders) | 4 (5) | 6 (6) | 2 (2)
58900-Obstruction gastric (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
59700-Oral pain (Gastrointestinal disorders) | 2 (2) | 5 (5) | 0 (0)
75600-Small intestinal mucositis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
75700-Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 3 (3) | 2 (2)
81900-Typhlitis (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1)
87900-Vomiting (Gastrointestinal disorders) | 7 (8) | 4 (4) | 8 (10)
28200-Edema face (General disorders) | 1 (1) | 0 (0) | 0 (0)
33200-Fatigue (General disorders) | 1 (1) | 0 (0) | 1 (1)
33900-Fever (General disorders) | 4 (4) | 1 (1) | 1 (1)
37200-General disorders and administration site conditions - Other specify (General disorders) | 1 (1) | 0 (0) | 0 (0)
48700-Irritability (General disorders) | 1 (1) | 0 (0) | 0 (0)
60600-Pain (General disorders) | 1 (1) | 0 (0) | 4 (4)
35500-Gallbladder pain (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
40600-Hepatobiliary disorders - Other specify (Hepatobiliary disorders) | 2 (2) | 2 (2) | 1 (1)
66500-Portal hypertension (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
12000-Allergic reaction (Immune system disorders) | 0 (0) | 1 (2) | 0 (0)
13100-Anaphylaxis (Immune system disorders) | 0 (0) | 2 (2) | 1 (1)
44700-Immune system disorders - Other specify (Immune system disorders) | 0 (0) | 1 (1) | 1 (1)
13400-Anorectal infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
16800-Bladder infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
20500-Catheter related infection (Infections and infestations) | 6 (7) | 5 (5) | 4 (4)
25600-Device related infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
29500-Enterocolitis infectious (Infections and infestations) | 4 (4) | 2 (2) | 4 (4)
38300-Gum infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
44800-Infections and infestations - Other specify (Infections and infestations) | 36 (48) | 32 (45) | 39 (68)
53100-Lung infection (Infections and infestations) | 4 (4) | 1 (1) | 2 (2)
60100-Otitis media (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
62500-Pelvic infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
66100-Pleural infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
73700-Sepsis (Infections and infestations) | 16 (16) | 11 (13) | 2 (3)
75200-Skin infection (Infections and infestations) | 1 (1) | 2 (2) | 1 (1)
76000-Small intestine infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (2)
82300-Upper respiratory infection (Infections and infestations) | 2 (2) | 1 (1) | 1 (1)
83100-Urinary tract infection (Infections and infestations) | 0 (0) | 2 (2) | 2 (2)
88900-Wound infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
14500-Arterial injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
34900-Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
46500-Intraoperative arterial injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 3 (3)
66800-Postoperative hemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 3 (3)
66900-Postoperative thoracic procedure complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
80700-Tracheal obstruction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
86400-Vascular access complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
10900-Activated partial thromboplastin time prolonged (Investigations) | 0 (0) | 2 (2) | 1 (1)
11600-Alanine aminotransferase increased (Investigations) | 18 (18) | 12 (14) | 8 (9)
11800-Alkaline phosphatase increased (Investigations) | 1 (1) | 1 (1) | 0 (0)
15000-Aspartate aminotransferase increased (Investigations) | 19 (19) | 11 (11) | 7 (7)
17400-Blood bilirubin increased (Investigations) | 1 (1) | 2 (2) | 1 (2)
24100-Creatinine increased (Investigations) | 3 (3) | 2 (2) | 0 (0)
34000-Fibrinogen decreased (Investigations) | 1 (1) | 1 (1) | 3 (3)
37500-GGT increased (Investigations) | 3 (3) | 5 (5) | 1 (2)
45800-INR increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
52600-Lipase increased (Investigations) | 0 (0) | 1 (1) | 1 (1)
53700-Lymphocyte count decreased (Investigations) | 13 (17) | 11 (16) | 12 (16)
58300-Neutrophil count decreased (Investigations) | 185 (254) | 148 (192) | 217 (287)
65800-Platelet count decreased (Investigations) | 146 (237) | 124 (177) | 175 (269)
73900-Serum amylase increased (Investigations) | 0 (0) | 2 (2) | 1 (1)
83600-Urine output decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
88300-Weight loss (Investigations) | 2 (2) | 0 (0) | 0 (0)
88500-White blood cell decreased (Investigations) | 32 (48) | 30 (42) | 36 (52)
10700-Acidosis (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 1 (1)
11900-Alkalosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
13500-Anorexia (Metabolism and nutrition disorders) | 16 (21) | 13 (17) | 11 (16)
24700-Dehydration (Metabolism and nutrition disorders) | 4 (4) | 2 (2) | 7 (7)
41300-Hypercalcemia (Metabolism and nutrition disorders) | 4 (4) | 0 (0) | 2 (2)
41400-Hyperglycemia (Metabolism and nutrition disorders) | 8 (8) | 13 (15) | 11 (12)
41600-Hyperkalemia (Metabolism and nutrition disorders) | 7 (7) | 6 (6) | 2 (3)
41700-Hypermagnesemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
42500-Hyperuricemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
42600-Hypoalbuminemia (Metabolism and nutrition disorders) | 2 (2) | 2 (2) | 2 (3)
42700-Hypocalcemia (Metabolism and nutrition disorders) | 10 (10) | 12 (13) | 5 (7)
42900-Hypoglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
43100-Hypokalemia (Metabolism and nutrition disorders) | 38 (48) | 36 (43) | 22 (26)
43200-Hypomagnesemia (Metabolism and nutrition disorders) | 3 (3) | 1 (1) | 0 (0)
43300-Hyponatremia (Metabolism and nutrition disorders) | 6 (7) | 11 (13) | 8 (8)
43500-Hypophosphatemia (Metabolism and nutrition disorders) | 3 (3) | 2 (2) | 4 (4)
48500-Iron overload (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
14700-Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
16200-Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
37300-Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
55900-Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
60700-Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
58000-Neoplasms benign malignant and unspecified (incl cysts and polyps) - Other specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
15300-Ataxia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
22000-Cognitive disturbance (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
25300-Depressed level of consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
31800-Extrapyramidal disorder (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
38800-Headache (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
58100-Nervous system disorders - Other specify (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
63900-Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
64100-Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
73600-Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
11400-Agitation (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
23000-Confusion (Psychiatric disorders) | 0 (0) | 2 (2) | 0 (0)
11100-Acute kidney injury (Renal and urinary disorders) | 3 (3) | 1 (1) | 2 (2)
39300-Hematuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1)
62600-Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
11300-Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1) | 0 (0)
14100-Apnea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 1 (1)
15100-Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)
15400-Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
19200-Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
27800-Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 1 (1)
29700-Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 1 (1)
43900-Hypoxia (Respiratory, thoracic and mediastinal disorders) | 8 (11) | 3 (3) | 7 (7)
64900-Pharyngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
65300-Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
65900-Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 5 (5) | 4 (4)
66300-Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 1 (1)
68700-Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
69000-Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
71500-Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (2) | 0 (0)
71600-Respiratory thoracic and mediastinal disorders - Other specify (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 4 (4)
78100-Stridor (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
68400-Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
69700-Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0)
75300-Skin ulceration (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
84100-Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
42100-Hypertension (Vascular disorders) | 6 (6) | 1 (1) | 4 (5)
43600-Hypotension (Vascular disorders) | 9 (9) | 3 (3) | 5 (5)
53300-Lymph leakage (Vascular disorders) | 2 (2) | 0 (0) | 0 (0)
79600-Thromboembolic event (Vascular disorders) | 2 (3) | 0 (0) | 0 (0)
86500-Vascular disorders - Other specify (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
87500-Visceral arterial ischemia (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Must obtain prior Sponsor approval.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2011-08-16): https://cdn.clinicaltrials.gov/large-docs/67/NCT00567567/Prot_SAP_000.pdf